CLINICAL TRIAL: NCT07331415
Title: Evaluation of Lifestyle Education and Events Via Network Text Messages After Acute Coronary Syndrome (Elena Trial)
Brief Title: Evaluation of Lifestyle Education and Events Via Network Text Messages After Acute Coronary Syndrome
Acronym: Elena
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación EPIC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EPIC50-Elena Trial
Record Dates: First submitted 2025-12-28; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Acute Coronary Syndrome; Myocardial Infarction; Cardiovascular Diseases
Keywords: Text messaging; Usual care
MeSH Terms: conditions — Acute Coronary Syndrome; Myocardial Infarction; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Text messaging group with usual care (Experimental)
  Interventions: Other: Text messaging and Usual Care
- Usual Care (Active Comparator)
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Other: Text messaging and Usual Care — The patient received a monthly telephone text messages (TTM) for 12 months with the recommendations of the Spanish Society of Cardiology regarding secondary prevention and followed the usual review protocol in a specific ischemic heart disease consultation at 3 and 12 months after discharge.
  Arms: Text messaging group with usual care
Behavioral: Usual Care — The patient received followed the usual review protocol in a specific ischemic heart disease consultation at 3 and 12 months after discharge.
  Arms: Usual Care

SUMMARY:
To evaluate the usefulness of telephone text messages (TTM) in the control of risk factors and in the reduction of events in the first year after an ACS (acute coronary syndrome).

DETAILED DESCRIPTION:
To evaluate the usefulness of telephone text messages (TTM) in the control of risk factors and in the reduction of events in the first year after an ACS (acute coronary syndrome).

ELIGIBILITY:
Inclusion Criteria:

* Patients discharged with ACS and without ST elevation.
* Informed consent signed.

Exclusion Criteria:

* Refusal to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 370 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Composite of cardiac death, myocardial infarction, stroke or new revascularization | 12 months
  Occurrence of Composite of cardiac death, myocardial infarction, stroke or new revascularization

SECONDARY OUTCOMES:
Systolic blood pressure (SBP) mm Hg | 12 months
  Mean of SBP
Diastolic blood pressure (DBP) (mm Hg) | 12 months
  Mean of DBP
Change in Weight (kilograms) | 12 months
  Mean of Change in Weight
Low Density Lipoproteins (LDL) cholesterol (mg/dl) | 12 months
  Mean of LDL
High (HDL) cholesterol (mg/dl) | 12 months
  Mean of LDL
Triglycerides (mg/dl) | 12 months
  Mean of Triglycerides
Glycosylated hemoglobin (%) | 12 months
  Mean of Glycosylated hemoglobin
Active smoking | 12 months
  Percentage of Active smoking
Exercise per week (hours) | 12 months
  Mean of Exercise per week
Total Death | 12 months
  Occurrence of All Death
Cardiac Death | 12 months
  Occurrence of Cardiovascular Death
Myocardial Infarction | 12 months
  Occurrence of Myocardial Infarction
Stroke | 12 months
  Occurrence of Stroke
New revascularization | 12 month
  Occurrence of New revascularization

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario de Cabueñes, Cabueñes, Spain

REFERENCES:
- [Background] Free C, Phillips G, Galli L, Watson L, Felix L, Edwards P, Patel V, Haines A. The effectiveness of mobile-health technology-based health behaviour change or disease management interventions for health care consumers: a systematic review. PLoS Med. 2013;10(1):e1001362. doi: 10.1371/journal.pmed.1001362. Epub 2013 Jan 15. PMID 23349621
- [Background] Sharma P APMptm, in fpatat, en/ pwHiRchawirhacsc, 2015). aF.
- [Background] Anglada-Martinez H, Riu-Viladoms G, Martin-Conde M, Rovira-Illamola M, Sotoca-Momblona JM, Codina-Jane C. Does mHealth increase adherence to medication? Results of a systematic review. Int J Clin Pract. 2015 Jan;69(1):9-32. doi: 10.1111/ijcp.12582. Epub 2014 Dec 4. PMID 25472682
- [Background] Adler AJ, Casas JP, Martin N, Free C, Perel P. Cochrane corner: text messaging to improve adherence to drugs for secondary prevention of cardiovascular disease. Heart. 2018 Nov;104(22):1814-1816. doi: 10.1136/heartjnl-2017-312888. Epub 2018 May 14. No abstract available. PMID 29760242
- [Background] Senatore FF, Califf RM. Standardized classification and framework for reporting and interpreting medication non-adherence in clinical trials. Eur Heart J. 2019 Jul 1;40(25):2086-2088. doi: 10.1093/eurheartj/ehy759. No abstract available. PMID 30496403